CLINICAL TRIAL: NCT00742261
Title: An Open-label, Randomized, Two-way Balanced Crossover Study to Investigate the Bioavailability of Two Forms ofGSK1363089 in Subjects With Solid Tumors
Brief Title: A Bioavailability Study of GSK1363089 in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MET111516
Record Dates: First submitted 2008-08-26; First posted 2008-08-27 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Solid Tumours
Keywords: Pharmacokinetics; Safety; MET; Bioavailability; Patients; GSK1363089A; GSK1363089G; GSK1363089; Relative
MeSH Terms: interventions — GSK 1363089

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK1363089 (Experimental): Two-part study to evlauate the relative bioavailability of GSK1363089 from a free base formulation (GSK1363089G) compared with the biophosphate salt formulation (GSK1363089A) (Part 1) and to assess the safety of the GSK1363089 biophosphate formulation when administered three times a week until disease progression (Part 2).
  Interventions: Drug: GSK1363089

INTERVENTIONS:
Drug: GSK1363089 — Two-part study to evlauate the relative bioavailability of GSK1363089 from a free base formulation (GSK1363089G) compared with the biophosphate salt formulation (GSK1363089A) (Part 1) and to assess the safety of the GSK1363089 biophosphate formulation when administered three times a week until disease progression (Part 2).
  Other Names: GSK1363089G; GSK1363089A

SUMMARY:
Study to compare 2 different chemical forms of GSK1363089.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of solid tumor malignancy.
* 18 years old with ECOG of 0-1.
* female subject who is not pregnant
* Male subjects must agree to use contraception methods
* Able to swallow and retain oral medication.
* The subject will refrain from the use of illicit drugs and adhere to other protocol-stated restrictions while participating in the study.
* QTcB or QTcF < 470 msec.
* Bilirubin = 1.5mg/dl, AST, ALT, ALP <2X ULN in absence of malignant disease in the liver or <5X ULN in case of liver involvement by the tumor.
* Serum Creatinine <1.5mg/dL

Exclusion Inclusion:

* The subject has received anticancer treatment.
* The subject has participated in a clinical trial and has received an investigational product within 21 days.
* The subject has known brain metastases.
* The subject has uncontrolled intercurrent illness.
* History of sensitivity to any of the study medications, or components.
* The subject is known to be positive for the human immunodeficiency virus (HIV).
* Subjects who have had partial or complete gastrectomy.
* Pregnant females as determined by positive ß-hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-08-11 (Actual); Primary Completion 2009-06-24 (Actual); Study Completion 2009-06-24 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters,Cmax, AUC(0-t), AUC(0-8)] from free base and bisphosphate salt formulations in Part 1 of the study. | 12 months

SECONDARY OUTCOMES:
Safety and tolerability in Part 1 and 2.• Time to tmax and t½ of GSK1363089in Part 1.• Trough and nominal peak GSK1363089 concentrations during Week 3 of Part 2.• Assess response to therapy in Part 2 of the study. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Naing A, Kurzrock R, Adams LM, Kleha JF, Laubscher KH, Bonate PL, Weller S, Fitzgerald C, Xu Y, LoRusso PM. A comparison of the pharmacokinetics of the anticancer MET inhibitor foretinib free base tablet formulation to bisphosphate salt capsule formulation in patients with solid tumors. Invest New Drugs. 2012 Feb;30(1):327-34. doi: 10.1007/s10637-010-9536-x. Epub 2010 Sep 15. PMID 20842406
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study MET111516 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/MET111516?search=study&study_ids=111516#rs
- Available data/document: Dataset Specification: MET111516 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: MET111516 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: MET111516 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: MET111516 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: MET111516 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: MET111516 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: MET111516 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register